CLINICAL TRIAL: NCT04460794
Title: Feasibility of a Novel Ballet-inspired Low-impact At-home Workout Programme to Improve Balance, Gait and Memory in Adults with Stroke: a Mixed Methods Exploratory Trial
Brief Title: A Novel Ballet-inspired Low-impact At-home Workout Programme for Adults with Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Suzanne HS Lo, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: FBB
Record Dates: First submitted 2020-07-03; First posted 2020-07-08 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-02

CONDITIONS: Stroke; Gait, Unsteady; Balance; Distorted; Memory Impairment
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic; Memory Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ballet-inspired workout programme (Group A) (Experimental): Participants will continue their usual activities and exercises, and in addition, receive an 8-week home-based programme delivered by trained volunteers via hybrid on-site and virtual contacts, and supported by volunteer healthcare professionals. A self-directed resource package will be developed.
  Interventions: Behavioral: Ballet-inspired workouts
- Usual care (Group B) (Other): Control participants will continue their usual activities and exercises during the study period. In addition, they will be provided with an information sheet about recommendations with pictorial demonstrations on basic stretching and leg exercises for stroke survivors.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Ballet-inspired workouts — 8 weeks, delivered by volunteers with a self-directed resource package
  Arms: Ballet-inspired workout programme (Group A)
Other: Usual care — Usual care and general recommendations on basic stretching and leg exercises for stroke survivors
  Arms: Usual care (Group B)

SUMMARY:
To explore the feasibility of a novel ballet-inspired low-impact at-home workout programme for community-dwelling stroke survivors in Hong Kong.

DETAILED DESCRIPTION:
A mixed methods exploratory study incorporating a randomised controlled trial (RCT) and qualitative evaluation will be conducted. A total of 40 stroke participants will be recruited from two acute public hospitals. Participants will be randomly assigned to receive the interention and usual care, or usual care only. Data will be collected in multiple forms: recruitment/retention rates, adherence to the intervention, journals, field notes, verbal feedback, audio records, semi-structured interviews, and questionnaires on outcomes (balance, confidence in balance, gait, walking endurance). This study is the first of its kind in Hong Kong. Findings will address the cross-cultural applicability of dance interventions and lay the groundwork for examination in a larger-RCT about its effects on survivors' balance, gait and memory.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 years or above
2. clinically diagnosed with a first-ever ischaemic/ haemorrhagic stroke
3. living in home settings
4. mild-moderate lower limb paresis with a modified Functional Ambulation Classification (MFAC) of III (Dependent walker) or above
5. a Montreal Cognitive Assessment (MoCA) score>20
6. able to follow three-step directions
7. able to communicate in Cantonese and read Traditional Chinese
8. their hearing and/or visual disturbances corrected by hearing aids and/or glasses
9. consent to participate in the study

Exclusion Criteria:

1. diagnosed with transcient ischaemic attack, subdural or epidural haemorrhage
2. experienced cerebrovascular events due to tumours or head trauma
3. have pre-existing neurological, cardiovascular or orthopaedic conditions that contradict participation in dancing such as shoulder dislocation, myocardial infarction, seizures or acutes illness
4. mental condition such as depression, schizophrenia or personality disorder
5. incomprehensible speech
6. severe hearing and/or visual disturbance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in the participants' level of balance | Change from baseline to immediately after completion of the intervention (over 8 weeks)
  The 14-item Mini-Balance Evaluation Systems Test (Mini-BESTest) will be used. It measures four domains: anticipatory postural adjustments, reactive postural control, sensory orientation, dynamic gait. Items are rated on a 3-level scale (0="Severe", 1="Moderate", 2="Normal"). Summed total score=0-28 (higher scores representing better balance ability). Cronbach alpha=0.89-0.94.

SECONDARY OUTCOMES:
Change in the participants' level of balance confidence | Change from baseline to immediately after completion of the intervention (over 8 weeks)
  The 16-item Activities-specific Balance Confidence Scale (Chinese version) will be adopted. Participants will rate their confidence in balance associated with performing 16 daily functional activities from 0% (absolutely no confidence) to 100% (fully confident). Summed total score=0-100% (higher scores denotes higher confidence). Cronbach alpha=0.97.
Change in the participants' level of gait | Change from baseline to immediately after completion of the intervention (over 8 weeks)
  The 31-item Gait Assessment and Intervention tool (G.A.I.T.) will be used to measure gait: upper extremity and trunk movement control; trunk and lower extremity (stance phase); trunk and lower extremity (swing phase). Each item is scored from 0 (normal) to 3, with gradients of variation from normal (Total score: 0 (normal gait) to 62 (greatest extent of gait deviations)). It has good intra-rater and interrater reliability.
Change in participants' level of walking endurance | Change from baseline to immediately after completion of the intervention (over 8 weeks)
  The 6-Minute Walk Test (MWT) will be performed in accordance with American Thoracic Society guidelines. The distance walked, the time stopped and reason(s) for stopping prematurely will be recorded. 6MWT, 12MWT, and self-paced gait speed were all significantly highly correlated (r>0.90).
Change in participants' level of memory | Change from baseline to immediately after completion of the intervention (over 8 weeks)
  The 11-item Rivermead Behavioural Memory Test - Third Version (Chinese version) will be used. For each task, scores range from 0-2 (2-points=normal; 1-point=intermediate; 0-point=error). Total score=0-254. It demonstrated a high inter-rater reliability. Correlation between performance on parallel forms=0.67-0.84.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Lo, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Alice Ho Miu Ling Nethersole Hospital, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analysed during the current study will be available from the corresponding author on reasonable request.
Supporting Information: Study Protocol
Time Frame: The datasets used and/or analysed during the current study will be available from the corresponding author on reasonable request, for six years upon completion of the study.
Access Criteria: The datasets used and/or analysed during the current study will be available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Lo SHS, Chau JPC, Choi KC, Yeung J, Li SH, Demers M. Feasibility of a ballet-inspired low-impact at-home workout programme for adults with stroke: a mixed-methods exploratory study protocol. BMJ Open. 2021 Apr 13;11(4):e045064. doi: 10.1136/bmjopen-2020-045064. PMID 33849853